CLINICAL TRIAL: NCT07319793
Title: Clinical Study on Optimized Treatment for Allogeneic Hematopoietic Stem Cell Transplantation in Relapsed/Refractory Myeloid Neoplasms
Brief Title: Pre-DLI or Pro-DLI in Relapsed/Refractory Myeloid Neoplasms After HSCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Chief, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-z240
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes (MDS)
Keywords: Donor lymphocyte infusion, DLI; Relapsed and refractory, R/R; myeloid neoplasms, MN
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic DLI (Experimental): DLI is performed between day +45 and day +60 post-transplantation. Peripheral blood hematopoietic stem cells are infused, with short-course immunosuppressive therapy administered after DLI. The infused mononuclear cell and CD3⁺ cell doses are 1.0×10⁸/kg and 3.0×10⁷/kg, respectively. Following DLI, graft-versus-host disease (GVHD) prophylaxis is administered using cyclosporine A or methotrexate. For patients undergoing fully matched transplants, prophylaxis lasts 4-6 weeks; for those receiving haploidentical transplants, it lasts 6-8 weeks.
  Interventions: Other: Prophylactic DLI
- Preemptive DLI (Active Comparator): DLI is initiated if the patient meets the criteria for MRD positivity. The regimen includes chemotherapy followed by DLI. Chemotherapy is administered 48-72 hours prior to peripheral blood hematopoietic stem cell infusion, using one of the following regimens: HAA (homoharringtonine + aclarubicin + cytarabine), AA (aclarubicin + cytarabine), HA (homoharringtonine + cytarabine), or VA (venetoclax + azacitidine). The principles of cell infusion and subsequent short-course immunosuppressive therapy are the same as in the prophylactic DLI group.
  Interventions: Other: Preemptive DLI

INTERVENTIONS:
Other: Prophylactic DLI — DLI is performed between day +45 and day +60 post-transplantation. Peripheral blood hematopoietic stem cells are infused, with short-course immunosuppressive therapy administered after DLI. The infused mononuclear cell and CD3⁺ cell doses are 1.0×10⁸/kg and 3.0×10⁷/kg, respectively. Following DLI, graft-versus-host disease (GVHD) prophylaxis is administered using cyclosporine A or methotrexate. For patients undergoing fully matched transplants, prophylaxis lasts 4-6 weeks; for those receiving haploidentical transplants, it lasts 6-8 weeks.
  Arms: Prophylactic DLI
Other: Preemptive DLI — DLI is initiated if the patient meets the criteria for MRD positivity. The regimen includes chemotherapy followed by DLI. Chemotherapy is administered 48-72 hours prior to peripheral blood hematopoietic stem cell infusion, using one of the following regimens: HAA (homoharringtonine + aclarubicin + cytarabine), AA (aclarubicin + cytarabine), HA (homoharringtonine + cytarabine), or VA (venetoclax + azacitidine). The principles of cell infusion and subsequent short-course immunosuppressive therapy are the same as in the prophylactic DLI group.
  Arms: Preemptive DLI

SUMMARY:
Donor lymphocyte infusion (DLI) based on minimal residual disease (MRD) has been widely adopted worldwide to enhance the graft-versus-leukemia effect following allogeneic hematopoietic stem cell transplantation (allo-HSCT). However, there is a lack of studies comparing the efficacy and safety of prophylactic versus preemptive DLI in patients with refractory/relapsed (R/R) acute myeloid leukemia (AML), and its effectiveness in other myeloid neoplasms (MN, such as myelodysplastic syndromes with excess blasts, MDS-IB) remains unknown, particularly with a scarcity of data from randomized controlled trials. This multicenter, randomized controlled study aims to prospectively compare the efficacy and safety of prophylactic versus preemptive DLI in patients with R/R myeloid neoplasms undergoing allo-HSCT. The study will enroll patients with MN (including AML and MDS-IB, excluding Ph+ cases) undergoing allo-HSCT, who are in R/R status at the time of transplant and achieve MRD-negative remission at 1 month post-transplant. Eligible patients must have no evidence of graft-versus-host disease (GVHD) or controlled GVHD, no severe infections, and no organ failure within 30-60 days post-transplant. One hundred patients will be enrolled in both the experimental and control groups. The primary endpoint is the relapse rate at 1 year post-randomization. Secondary endpoints include: 1-year leukemia-free survival and overall survival, and the incidence of bone marrow suppression, pancytopenia, GVHD, and infections following DLI. This study aims to explore strategies to reduce relapse rates and improve survival in patients with R/R MN following allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were those who underwent allogeneic hematopoietic stem cell transplantation (allo-HSCT) for myeloid neoplasms (MN), excluding Philadelphia chromosome-positive (Ph+) disease, regardless of age. MN included acute myeloid leukemia (AML) and myelodysplastic syndrome with increased blasts (MDS-IB). Patients were required to have refractory or relapsed disease at the time of transplantation, defined as >5% blasts in the bone marrow after salvage chemotherapy and prior to the transplant conditioning regimen. Additionally, patients must have achieved minimal residual disease (MRD)-negative remission within 1 month post-transplantation. All participants provided voluntary written informed consent.

Exclusion Criteria:

* Early mortality or relapse within 30 days post-transplantation.
* Active graft-versus-host disease (GVHD) not under control between 30 and 60 days post-transplantation.
* Presence of severe or uncontrolled infections.
* Presence of significant organ dysfunction, defined as:

Hepatic dysfunction: Known severe cirrhosis, portal hypertension, or active liver disease; or laboratory-confirmed alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3.0 × the upper limit of normal (ULN) and/or total bilirubin (TBIL) > 1.5 × ULN.

Renal dysfunction: Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m² (calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation) or serum creatinine > 1.5 × ULN; or requirement for regular hemodialysis or peritoneal dialysis.

Cardiac dysfunction: New York Heart Association (NYHA) functional class III or IV; unstable angina, acute myocardial infarction, coronary artery bypass grafting (CABG), or percutaneous coronary intervention (PCI) within 6 months prior to enrollment; left ventricular ejection fraction (LVEF) < 50% (confirmed by echocardiography or other Doppler examination); clinically significant, uncontrolled arrhythmia.

Respiratory dysfunction: Chronic obstructive pulmonary disease (COPD) or other pulmonary disease requiring long-term oxygen therapy; resting oxygen saturation (SpO₂) < 92% on room air.

* Participation in another investigational drug trial within the 3 months prior to enrollment.
* Any other condition deemed by the investigator to make the patient unsuitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Relapse | From study enrollment until the 1-year follow-up
  The cumulative incidence of relapse at 1 year post-randomization.

SECONDARY OUTCOMES:
LFS | From study enrollment until the 1-year follow-up
  1 year leukemia-free survival
OS | From study enrollment until the 1-year follow-up
  1-year overall survival
Incidence of bone marrow suppression | From study enrollment until the 1-year follow-up
  Incidence of bone marrow suppression, including neutropenia, anemia, thrombocytopenia, and pancytopenia
GVHD | From study enrollment until the 1-year follow-up
  1-year acute and chronic graft-versus-host disease
Infection | From study enrollment until the 1-year follow-up
  1-year incidence of infections (bacterial, viral, and fungal)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided